CLINICAL TRIAL: NCT01239680
Title: Biological Response of Trauma Patients to Standard Trauma Resuscitation Therapy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-18
Record Dates: First submitted 2010-10-12; First posted 2010-11-11 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Hemorrhagic Shock
Keywords: hemorrhagic shock; glutamine; trauma resuscitation; department of defense; trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries | interventions — Glutamine; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ringer's Lactate and Placebo for Glutamine (Placebo Comparator): Ringer's Lactate 1 liter once over 6 hours
  Interventions: Drug: Ringer's Lactate; Drug: Placebo (for Glutamine)
- Ringer's Lactate with 25 grams Glutamine (Experimental): Ringer's Lactate with 25 grams Glutamine (1 liter) once over 6 hours
  Interventions: Drug: Glutamine; Drug: Ringer's Lactate

INTERVENTIONS:
Drug: Glutamine — Intravenous 25 grams once over 6 hours
  Arms: Ringer's Lactate with 25 grams Glutamine
Drug: Ringer's Lactate — Intravenous 1 liter once over 6 hours
  Other Names: Lactated Rigner's (LR)
Drug: Placebo (for Glutamine) — Given Intravenously in 1 liter Lactated Ringer's
  Arms: Ringer's Lactate and Placebo for Glutamine

SUMMARY:
Overall aim of this work is to evaluate new methods of resuscitation that can be applied by front-line responders on the battlefield, in civilian life, or which can be used during initial resuscitation in the first fixed facility to which the injured patient is brought.

DETAILED DESCRIPTION:
Shock is a leading cause of death among American forces in battle, with many trauma victims dying of early hemorrhagic shock or from late septic shock.1 Shock is defined as circulatory collapse, when the arterial blood pressure is too low to maintain an adequate supply of blood to the body's vital organs and tissues. Specifically, hemorrhagic shock results when blood vessels are physically damaged while septic shock results when microbes or microbial products enter the blood stream. Despite advances in medical science, including the development of improved antibiotics, treatments for hemorrhagic and septic shock have changed little in the past 30-40 years. A wounded soldier bleeding on the battlefield, or a trauma victim in the United States, is treated today largely as he or she would have been treated in 1970.

The overall aim of this work is to evaluate new methods of resuscitation that can be applied by front-line responders on the battlefield (medical corpsmen, combat medics), in civilian life (Emergency Medical System), or which can be used during initial resuscitation in the first fixed facility to which the injured patient is brought. This might be a Fire Support Specialist (FIST) team in a combat theater or a trauma center in the civilian health care system.

ELIGIBILITY:
Inclusion Criteria:

* Blunt or penetrating trauma patients who meet Truman Medical Center criteria for a trauma activation.
* These patients will typically be in shock and have blunt injuries or penetrating trauma.
* Patients must be alert, awake, oriented, and responsive and be English speaking males or females between the ages 21-65.

Exclusion Criteria:

* traumatic cardiac arrest patients,
* pregnant patients,
* interhospital transfer patients,
* non-English speaking patients,
* patients with suspected or confirmed Human Immunodeficiency Virus (HIV) or AIDs based on clear history,
* prior laboratory tests, or strong clinical suspicion; patients with clinical evidence of impaired mental function;
* patients with continuing hypotension or tachycardia after resuscitation;
* patients with blood alcohol in excess of 80mg/dl;
* signs suggestive of coagulopathy;
* allergy to glutamine;
* liver disease or renal disease.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Van Way, III, M.D., Principal Investigator — University of Missouri, Kansas City
Locations (2):
- United States (2):
  - Truman Medical Center-Hospital Hill, Kansas City, Missouri
  - Univeristy of Missouri-Kansas City, Kansas City, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period started 01/12/2011. Recruitment ended 11/01/2013. Subjects were recruited from the Emergency Department and Intensive Care Units at Truman Medical Center Hospital Hill. These subjects were Trauma Activations. Recruitment was performed by the Principal Investigator, Research Coordinator, or other approved study staff.
Groups:
- Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours: Administration of Ringer's Lactate per Advanced Trauma Life Support Protocol with additional Ringer's Lactate: Ringer's Lactate Intravenous 1 liter once over 6 hours
- Glutamine: Intravenous 25 Grams Once Over 6 Hours: Administration of Ringer's Lactate per Advanced Trauma Life Support Protocol with additional glutamine: Glutamine: Intravenous 25 grams once over 6 hours
Period: Overall Study
Arm/Group | Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours | Glutamine: Intravenous 25 Grams Once Over 6 Hours
Started | 3 | 2
Completed | 1 | 2
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours: Administration of Ringer's Lactate per Advanced Trauma Life Support Protocol with additional Ringer's Lactate: Ringer's Lactate: Intravenous 1 liter once over 6 hours
- Total: Total of all reporting groups
Arm/Group | Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours | Glutamine: Intravenous 25 Grams Once Over 6 Hours | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Customized [Number; unit: participants] — Age 21 to 65 years.
  participants
    Age 21-65 | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Biological Response as Characterized by Selected Cytokines, Specifically Tumor Necrosis Factor Alpha (TNFα), Interleukin One (IL-1β), and Interleukin Six (IL-6).
Description: Biological response as characterized by selected cytokines, specifically tumor necrosis factor alpha (TNFα), interleukin one (IL-1β), and interleukin six (IL-6). These are measured using ELISA. Baseline values are expected to be either unobtainable, or in any case less than 50 picograms/ml. If there is a significant inflammatory response, values at 24 hours should be more than 100 picograms/ml for TNFα, IL-1β, and IL-6. Our hypothesis is that there will be a difference between study and control group patients of at least 50 picograms/ml in the levels of these cytokines at 24 hours. Cytokine response is quite variable, and the percentage of outliers (with no cytokine response) in either group may be as high as 50%. .
Time Frame: Change from Baseline in Cytokine Levels at 24 hours
Population: The number of participants who had an intervention and completed the study with all 3 required blood draws.
Arm/Group | Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours | Glutamine: Intravenous 25 Grams Once Over 6 Hours
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years total.
Description: Each study subjects was followed and assessed for Adverse events while enrolled in the study.
Arm/Group | Ringer's Lactate: Intravenous 1 Liter Once Over 6 Hours | Glutamine: Intravenous 25 Grams Once Over 6 Hours
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/3 | 0/2

LIMITATIONS AND CAVEATS:
Many subjects excluded due to being unstable after initial resuscitation, having altered mental status, inability to speak English, <21 years of age, or blood alcohol in excess of 80mg/dl. No waiver of consent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No